CLINICAL TRIAL: NCT04250311
Title: A Multicenter, Placebo-controlled, Double-blind, Randomized Clinical Trial in Parallel Groups to Evaluate the Efficacy and Safety of ММН-407 in the Treatment of Influenza in Outpatient Adults
Brief Title: Clinical Trial of Efficacy and Safety of ММН-407 in the Treatment of Influenza in Outpatient Adults
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to the end of the ARVI and influenza season, it was suspended until approximately October 01, 2023
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMH-407-002
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MMH-407 (Experimental): Oral administration. Single dose: 1 tablet. First 24 hours of therapy: 1 tablet every 30 minutes for the first 2 hours, followed by 3 more tablets taken at regular intervals during the rest of the day. Days 2 to 5: 1 tablet 3 times daily.
  Interventions: Drug: MMH-407
- Placebo (Placebo Comparator): Oral administration. Single dose: 1 tablet. First 24 hours of therapy: 1 tablet every 30 minutes for the first 2 hours, followed by 3 more tablets taken at regular intervals during the rest of the day. Days 2 to 5: 1 tablet 3 times daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MMH-407 — MMH-407: For oral use.
  Other Names: Raphamin
  Arms: MMH-407
Drug: Placebo — Placebo: For oral use.
  Arms: Placebo

SUMMARY:
The main purpose of this study is:

• to evaluate the efficacy and safety of MMH-407 in the treatment of influenza in outpatient adults.

DETAILED DESCRIPTION:
Design: a multicenter, placebo-controlled, double-blind, randomized clinical trial in parallel groups.

The study will include both male and female patients aged 18-64 years with clinical signs of influenza within the first 24 hours of the onset of illness.

The influenza diagnosis must be supported by a positive rapid test (detection of influenza virus antigens in nasal epithelial cells). After the patients provide signed Participant Information Sheet and Informed Consent form, their medical history and body temperature will be recorded and physical examination and rapid diagnostic test performed. Patients who test positive will be assessed for 7 influenza-associated symptoms: cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, fatigue.

4-point Flu Symptom Severity scale will be used: 0 = no symptom; 1 = mild symptom; 2 = moderate symptom; 3 = severe symptom.

Nasopharyngeal swabs will be obtained from these patients for subsequent real-time reverse transcription polymerase chain reaction (RT-PCR) influenza A/B testing and laboratory tests performed.

If a patient meets all inclusion criteria and does not meet any of the exclusion criteria at Visit 1 (Day 1), he/she will be randomized into one of the treatment groups: Group 1: ММН-407 for 5 days, or Group 2: Placebo on the ММН-407 regimen for 5 days.

The patients will use electronic patient diaries to daily record their morning and evening axillary temperature (taken using a Geratherm mercury-free thermometer) and severity of 7 influenza-associated symptoms (using the Flu Symptom Severity scale). In addition to this, the patients will record doses of antipyretic drugs taken (when applicable) and any worsening of their health status (when applicable, to assess treatment safety and collect adverse events data).

In total, patients will be observed for 14 days (screening and randomization - up to 24 hours, treatment - 5 days, subsequent observation - up to 2 days; and a follow-up 'telephone' visit - Day 14).

During the study, 3 visits from patient to the physician's office and a follow-up telephone visit will be accomplished: 1) patient visits - Days 1, 3 and 7 (Visits 1, 2, and 3) at the medical centre; 2) telephone visit from the physician (Visit 4) - Day 14.

During Visits 2 and 3, the physician will perform a physical examination, record the changes in patients' symptoms and the use of concomitant medications and check the completion of patient diaries. At Visit 2, nasopharyngeal swabs for RT-PCR will be collected. Visit 3 will involve an assessment of treatment compliance and laboratory tests. The telephone visit is intended to provide information on a patient's health status, presence/absence of secondary bacterial complications and the use of antibiotics.

During the study, subjects will be allowed to use symptomatic therapy and medications for their co-morbidities, except for the medicines listed in the "Prohibited Concomitant Medications" section.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of male and female gender aged 18 to 64 years.
2. Uncomplicated, moderate influenza supported by all the symptoms:

   * axillary temperature ≥38.1°С on physician examination;
   * at least one moderate general symptom of influenza infection (headache, fever/chill, aches in the muscles/joints, weakness/drowsiness);
   * at least one moderate respiratory symptom of influenza infection (cough, sore throat, or nasal congestion).
3. Positive influenza rapid test (detection of virus antigens in the nasal epithelium).
4. First 24 hours of the onset of illness.
5. Patients who agree to use a reliable method of birth control during the study.
6. Patients who have provided signed Participant Information Sheet and Informed Consent form to participate in a clinical trial.

Exclusion Criteria:

1. Severe influenza infection that requires hospitalization.
2. Suspected pneumonia or bacterial infection (including otitis media, sinusitis, urinary tract infection, meningitis, sepsis, etc.) that requires the use of antibiotics, starting from the first day of illness.
3. Suspected early manifestations of a condition that, on its first onset, produces symptoms similar to those of influenza (other infectious diseases and/or influenza-like syndrome associated with the first onset of a systemic connective tissue disorder or another condition).
4. Patients who require the use of antivirals that are not permitted during the study.
5. Current season influenza vaccination.
6. Prior history or diagnosis of primary or secondary immunodeficiency
7. Patients with any known or suspected malignant neoplasm.
8. An exacerbated or decompensated chronic disease interfering with the subject's participation in the clinical trial.
9. Malabsorption syndrome, including congenital or acquired lactase deficiency (or any other disaccharidase deficiency), and/or galactosemia.
10. Current allergy to or intolerance of the active substances or any of the excipients in the medications used in the treatment.
11. Pregnancy, breast-feeding, childbirth within less than 3 months prior to the inclusion in the trial, or unwillingness to use contraceptive methods during the study
12. Prior history of non-adherence to medication; mental disorder; or alcohol or substance abuse, which, in the investigator's opinion, will compromise compliance with study procedures.
13. Use of any of the "Prohibited Concomitant Medications" within 2 weeks prior to study entry.
14. Patients who, as judged by the investigator, will fail or be unwilling to comply with the observation requirements or adhere to the dosing regimen during the study.
15. Participation in other clinical studies within 3 months prior to the inclusion in this study.
16. Patients who are related to any of the on-site research personnel directly involved in the conduct of the study or are an immediate relative of the investigator. 'Immediate relative' means husband, wife, parent, son, daughter, brother, or sister (regardless of whether they are natural or adopted).
17. Patients who work for OOO "NPF "Materia Medica Holding" (i.e. company employees, temporary contract workers, designated officials responsible for carrying out the research or any immediate relatives of the aforementioned).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 314 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Time to improvement of influenza symptoms. | On days 1-14 of observation.
  Based on patient diaries. In the morning and in the evening, the patients rate the severity of their symptoms on a 4-point scale (7 symptoms of influenza): headache, fever/chill, aches in the muscles/joints, weakness/drowsiness, cough, sore throat, and nasal congestion, where the absence of symptoms is 0, mild symptoms - 1, moderate symptoms - 2, and severe symptoms is 4. "Improvement of influenza symptoms" means no or mild symptoms.

SECONDARY OUTCOMES:
Proportion of patients reporting improvement of influenza symptoms. | On days 1-14 of observation period.
  Based on patient diaries.
Severity of illness. | On days 1- 6 of the observation period.
  Total symptom score AUC (to be estimated from each of the seven symptom subscores).
Proportion of patients with negative virus shedding. | On day 3 of the observation period.
  Negative influenza RT-PCR on nasopharyngeal swabs.
Dosing frequency of antipyretics according to indications. | On days 1-3 of the treatment period.
  A decrease dosing frequency of antipyretics while taking MMN-407 is one of the criteria for effectiveness. Based on patient diaries.
Proportion of subjects reporting worsening of illness. | On days 4 -14 of the observation period.
  Worsening of illness is bacterial complication of influenza that require the use of antibiotics or hospitalization.
Occurrence and nature of adverse events (AE). | On days 1-5 of the treatment period.
  AE severity, causal relationship to the study drug and outcome.
Number of patients with treatment-related changes in vital signs: body temperature, pulse rate (heart rate), respiration rate (breathing rate), and blood pressure. | On days 1- 5 of the treatment period.
  Based on medical records. Vital signs will be measured in a medical setting.
Proportion of subjects with clinically significant abnormal laboratory data. | On days 1- 5 of the treatment period.
  Вased on medical records.

CONTACTS AND LOCATIONS:
Locations (20):
- Russia (20):
  - Altai State Medical University, Department of Faculty Therapy with a course of immunology and allergology, Barnaul, Moscow
  - City Hospital # 5, Barnaul
  - Belgorod State National Research University, Hospital Therapy Department, Belgorod
  - Road Clinical Hospital at Chelyabinsk station of JSC Russian Railways, Chelyabinsk
  - City Clinical Hospital # 9 of the Ministry of Health of the Udmurt Republic, Izhevsk
  - Kazan State Medical University, Internal Medicine Department, Kazan'
  - Kuban State Medical University, Infectious Diseases and Phthisiopulmonology Department, Krasnodar
  - Central Clinical Hospital of the Russian Academy of Sciences, Moscow
  - City Clinical Hospital # 10 of the Kanavinsky District of Nizhny Novgorod, Nizhny Novgorod
  - Road Clinical Hospital at the station Nizhny Novgorod of JSC Russian Railways, Nizhny Novgorod
  - Vvedensky City Clinical Hospital, Saint Petersburg
  - City Polyclinic # 25 of the Nevsky District, Saint Petersburg
  - Medical Center "Reavita Med SPb", Saint Petersburg
  - Llc "Medical Clinic", Saint Petersburg
  - City Polyclinic # 43, Saint Petersburg
  - Samara City Hospital # 4, Samara
  - Scientific Medical Center for General Therapy and Pharmacology, Stavropol
  - Tver State Medical University, Department of Hospital Therapy, Tver'
  - Bashkir State Medical University, Internal Medicine Department, Ufa
  - Volgograd State Medical University, Volgograd